CLINICAL TRIAL: NCT03606980
Title: Iontophoresis With Dexamethasone in Combination With Physical Therapy for the Treatment of Pediatric Patients Diagnosed With Apophysitis of the Knee: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Iontophoresis With Dexamethasone and Physical Therapy to Treat Apophysitis of the Knee in Pediatrics
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Children's Health System, Inc. (Other)
Responsible Party: Principal Investigator, Dana Reesman, DPT, CHKD Sports Medicine Physical Therapist, Children's Health System, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHKDSM-001
Record Dates: First submitted 2018-06-29; First posted 2018-07-31 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Apophysitis; Juvenile
MeSH Terms: interventions — dexamethasone 21-phosphate; Iontophoresis; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Iontophoresis with Dexamethasone (Experimental): Iontophoresis is a non-invasive delivery mechanism for transmitting a medication to a local area of the body. The I-Bresis™ System and I-Bresis™ Patch will be the delivery system used for this study. The I-Bresis™ Patch is an adhesive patch. 1.5 ml of the dexamethasone sodium phosphate (4ml/1mL) will be placed on one side and 1.5 ml of 0.9% sodium chloride (saline) solution will be placed on the other. Duration of exposure: 123 minutes. Frequency of exposure: twice per week for a total of 12 sessions over a maximum of 8 weeks or until Return to Sport Criteria are met, whichever is sooner. Participants will also receive the standard PT protocol for apophysitis of the knee. This will involve up to 20 visits.
  Interventions: Drug: Dexamethasone Sodium Phosphate; Procedure: Iontophoresis; Procedure: Physical Therapy
- Iontophoresis with Sodium Chloride (Placebo Comparator): Iontophoresis is a non-invasive delivery mechanism for transmitting a medication to a local area of the body. The I-Bresis™ System and I-Bresis™ Patch will be the delivery system used for this study. The I-Bresis™ Patch is an adhesive patch. 1.5 ml of 0.9% sodium chloride (saline) solution will be placed on one side and 1.5 ml of 0.9% saline solution will be placed on the other. Duration of exposure: 123 minutes. Frequency of exposure: twice per week for a total of 12 sessions over a maximum of 8 weeks or until Return to Sport Criteria are met, whichever is sooner. Participants will also receive the standard PT protocol for apophysitis of the knee. This will involve up to 20 visits.
  Interventions: Procedure: Iontophoresis; Procedure: Physical Therapy
- Physical Therapy alone (Active Comparator): Participants will only receive the standard PT protocol for apophysitis of the knee. This will involve up to 20 visits.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate — Dexamethasone sodium phosphate administered via iontophoresis
  Arms: Iontophoresis with Dexamethasone
Procedure: Iontophoresis — Iontophoresis on affected knee
  Arms: Iontophoresis with Dexamethasone; Iontophoresis with Sodium Chloride
Procedure: Physical Therapy — Physical therapy of affected knee

SUMMARY:
The goal of this clinical research study is to determine if there is a difference in time to meet return to sport criteria for Pediatric patients with apophysitis of the knee who receive iontophoresis with Dexamethasone Sodium Phosphate (DSP) and Physical Therapy (PT) as those who receive iontophoresis with placebo and PT or PT alone.

Approximately 147 patients will be enrolled in this study.

DETAILED DESCRIPTION:
Iontophoresis is a treatment that allows medication to be delivered across your skin to the painful area without having to have an injection into your muscle or soft tissue, through a vein in your arm, or taking a pill. Instead, liquid medication is placed on a patch (like a large Band-Aid) and then placed on your knee over the location where it hurts. A plastic device, like a battery, is then attached to the patch for three minutes. During this time, this device begins to deliver the medication through your skin and into the area that hurts, and also charges the patch so it can continue to deliver the medication for two hours once the device is removed. The medication is delivered by a mild electrical current. The most common drug used with iontophoresis for pain caused by such things as apophysitis of the knee is dexamethasone sodium phosphate (dexamethasone).

This is an investigational study. Dexamethasone is a steroid medication that has been approved by the U.S Food and Drug Administration (FDA) to treat many types of problems (such as joint problems, skin and allergy problems, eye, stomach, and lung problems), but has not been approved to treat apophysitis of the knee using iontophoresis. In this study, it is an experimental drug.

Participants will be randomized to one of three treatment groups:

* Physical therapy with iontophoresis using Dexamethasone
* Physical therapy with iontophoresis using an inactive drug called a placebo
* Physical therapy alone

Participants will be asked to attend study visits twice/week for up to 8 weeks or until they are able to pass the Return To Sport Checklist, whichever is sooner. Participants will the receive a 30-Day Follow Up phone call and complete a survey at the 90-Day mark, making each participant's study duration approximately five (5) months.

ELIGIBILITY:
Inclusion Criteria:

1. Written approval from the referring physician for potential subject to be considered for enrollment into this study
2. Provision of signed and dated informed consent form
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. In good general health as evidenced by written approval from referring physician for potential inclusion in study.
5. Has the ability to effectively identify pain/burns and communicate with the investigators or their parents that they are experiencing pain or burning during treatment
6. Referred to CHKD Sports Medicine PT by CHKD Primary Care Sports Medicine physicians or CHKD Orthopedics physicians with a diagnosis of apophysitis of the knee and with a prescription for standard PT treatment with iontophoresis
7. Able and willing to complete iontophoresis treatments within eight (8) weeks of first treatment
8. Must be ambulatory
9. Males 7 to 14 years of age who have not reached skeletal maturity (skeletal maturity based on referring physician's clinical judgement or as demonstrated via radiograph images taken within 90 days of enrollment)
10. Females 7 to 14 years of age who have not reached skeletal maturity (skeletal maturity based on referring physician's clinical judgement or as demonstrated via radiograph images taken within 90 days of enrollment) and who meet one of the following criteria:

    1. Pre-menarcheal
    2. Within two (2) year post onset of menses
11. Males or females over the age of 14 only with radiographic evidence of skeletal immaturity, with images taken within 90 days of enrollment
12. Index knee symptomatic for pain with activities of daily living or while playing sports.

Exclusion Criteria:

1. Index knee symptomatic for pain only with palpation and not with activities of daily living or while playing sport
2. Diagnosis of bilateral apophysitis of the knee where both knees meet all of the inclusion criteria
3. Systemic fungal infections
4. Has an implanted electronic device
5. Has a known sensitivity to DSP
6. Presence of damaged skin, denuded skin, or other recent scar tissue on index knee
7. Presence of active dermatologic conditions in the affected area (e.g., eczema, psoriasis)
8. Presence of an abnormal neurological exam that indicates the subject would have a reduced ability to perceive pain (e.g. peripheral neuropathy)
9. Has a known sensitivity to electrical current
10. Is currently taking systemic steroids
11. Has had iontophoresis with DSP treatment within the past 30 days
12. Previously enrolled in this study
13. Currently enrolled in another treatment research study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Reesman, PT, DPT, Principal Investigator — Children's Hospital of the Kings Daughters
Locations (5):
- United States (5):
  - CHKD Sports Medicine Physical Therapy - Oakbrooke, Chesapeake, Virginia
  - CHKD Sports Medicine Physical Therapy - Tech Center, Newport News, Virginia
  - CHKD Sports Medicine Physicial Therapy - Ghent, Norfolk, Virginia
  - CHKD Sports Medicine Physical Therapy - Loehmann's Plaza, Virginia Beach, Virginia
  - CHKD Sports Medicine Physical Therapy - Landstown, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gholve PA, Scher DM, Khakharia S, Widmann RF, Green DW. Osgood Schlatter syndrome. Curr Opin Pediatr. 2007 Feb;19(1):44-50. doi: 10.1097/MOP.0b013e328013dbea. PMID 17224661
- [Background] Maffulli N, Longo UG, Spiezia F, Denaro V. Sports injuries in young athletes: long-term outcome and prevention strategies. Phys Sportsmed. 2010 Jun;38(2):29-34. doi: 10.3810/psm.2010.06.1780. PMID 20631461
- [Background] Circi E, Atalay Y, Beyzadeoglu T. Treatment of Osgood-Schlatter disease: review of the literature. Musculoskelet Surg. 2017 Dec;101(3):195-200. doi: 10.1007/s12306-017-0479-7. Epub 2017 Jun 7. PMID 28593576
- [Background] Kujala UM, Kvist M, Heinonen O. Osgood-Schlatter's disease in adolescent athletes. Retrospective study of incidence and duration. Am J Sports Med. 1985 Jul-Aug;13(4):236-41. doi: 10.1177/036354658501300404. PMID 4025675
- [Background] Joshi A, Stagni G, Cleary A, Patel K, Weiss DS, Hagins M. Iontophoresis successfully delivers dexamethasone sodium phosphate to dermis as measured by microdialysis. J Pharm Sci. 2014 Jan;103(1):191-6. doi: 10.1002/jps.23771. Epub 2013 Nov 6. PMID 24338751
- [Background] Nirschl RP, Rodin DM, Ochiai DH, Maartmann-Moe C; DEX-AHE-01-99 Study Group. Iontophoretic administration of dexamethasone sodium phosphate for acute epicondylitis. A randomized, double-blinded, placebo-controlled study. Am J Sports Med. 2003 Mar-Apr;31(2):189-95. doi: 10.1177/03635465030310020601. PMID 12642251
- [Background] Runeson L, Haker E. Iontophoresis with cortisone in the treatment of lateral epicondylalgia (tennis elbow)--a double-blind study. Scand J Med Sci Sports. 2002 Jun;12(3):136-42. doi: 10.1034/j.1600-0838.2002.02142.x. PMID 12135445
- [Background] Amirjani N, Ashworth NL, Watt MJ, Gordon T, Chan KM. Corticosteroid iontophoresis to treat carpal tunnel syndrome: a double-blind randomized controlled trial. Muscle Nerve. 2009 May;39(5):627-33. doi: 10.1002/mus.21300. PMID 19347928
- [Background] Neeter C, Thomee R, Silbernagel KG, Thomee P, Karlsson J. Iontophoresis with or without dexamethazone in the treatment of acute Achilles tendon pain. Scand J Med Sci Sports. 2003 Dec;13(6):376-82. doi: 10.1046/j.1600-0838.2003.00305.x. PMID 14617059
- [Background] Marovino T, Graves C. Iontophoresis in Pain Management. Practical Pain Management . 2011; 8(2): 1-2. Available from: https://www.practicalpainmanagement.com/treatments/interventional/iontophoresis-pain-management, Accessed May 17, 2018
- [Background] Dexamethasone sodium phosphate. In: Micromedex Solutions DRUGDEX® System. IBM Watson Health. Ann Arbor, MI. [cited April 22, 2018]. Available from: http://micromedexsolutions.com
- [Background] Dhote V, Bhatnagar P, Mishra PK, Mahajan SC, Mishra DK. Iontophoresis: a potential emergence of a transdermal drug delivery system. Sci Pharm. 2012 Jan-Mar;80(1):1-28. doi: 10.3797/scipharm.1108-20. Epub 2011 Dec 13. PMID 22396901
- [Background] Kaur J, Malik M, Sharma P, Sangwan P, Rani M. Effect of iontophoresis with dexamethasone in pain. Indian Journal of Physiotherapy and Occupational Therapy. 2017; 11(3).
- [Background] Clijsen R, Taeymans J, Baeyens JP, Barl AO, Clarys P. The effects of iontophoresis in the treatment of musculoskeletal disorders - a systematic review and meta-analysis. Drug Delivery Letters. 2012: 2(3).
- [Background] Goyal M, Kumar A, Mahajan N, Moitra M. Treatment of plantar fasciitis by taping vs. iontophoresis: a randomized clinical trial. Journal of Exercise Science and Physiotherapy. 2013: 9(1):34-39
- [Background] Mina R, Melson P, Powell S, Rao M, Hinze C, Passo M, Graham TB, Brunner HI. Effectiveness of dexamethasone iontophoresis for temporomandibular joint involvement in juvenile idiopathic arthritis. Arthritis Care Res (Hoboken). 2011 Nov;63(11):1511-6. doi: 10.1002/acr.20600. PMID 22034112
- [Background] Stefanou A, Marshall N, Holdan W, Siddiqui A. A randomized study comparing corticosteroid injection to corticosteroid iontophoresis for lateral epicondylitis. J Hand Surg Am. 2012 Jan;37(1):104-9. doi: 10.1016/j.jhsa.2011.10.005. PMID 22196293
- [Background] Vaishya R, Azizi AT, Agarwal AK, Vijay V. Apophysitis of the Tibial Tuberosity (Osgood-Schlatter Disease): A Review. Cureus. 2016 Sep 13;8(9):e780. doi: 10.7759/cureus.780. PMID 27752406
- [Background] WHO Physical activity and young people [Internet]. World Health Organization; c2018 [cited 2018 June 20]. Available from: http://www.who.int/dietphysicalactivity/factsheet_young_people/en/
- [Background] WHO Physical activity [Internet]. World Health Organization; c2018 [cited 2018 June 20]. Available from: http://www.who.int/dietphysicalactivity/pa/en/
- [Background] I-Bresis™ Charging Station (1360) - Instructions For Use [Internet]. Rev. B 2017 [cited 2018 May 17]. Available from: http://www.djoglobal.com/sites/default/files/Charging%20Station%20IFU.pdf
- [Background] I-Bresis™ Controller (1361) - Instructions For Use, [Internet]. Rev. B 2017 [cited 2018 May 17]. Available from: http://www.djoglobal.com/sites/default/files/Controller%20IFU.pdf
- [Background] I-Bresis™ Patch (5000060) - Instructions For Use, [Internet]. Rev. B 2017 [cited 2018 May 17]. Available from: http://www.djoglobal.com/sites/default/files/Electrode%20IFU.pdf
- [Background] Sodium Chloride Injection, USP [package insert]. Deerfield, IL: Baxter Corporation; 2018 [cited 2018 April 25]. Available from http://baxterpi.com/pi-pdf/Sodium_Chloride_Injection_Viaflex_PI.pdf
- [Background] 2007 Standard Operating Procedures of the Eastern Virginia Medical School Institutional Review Board [Internet]. July 2007 [cited 2018 May 17]. Available from: https://www.evms.edu/media/evms_public/departments/research_administration/research_subjects_protections/2007_EVMS_IRB_SOPs.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
Started | 16 | 15 | 14
Completed | 12 | 13 | 7
Not Completed | 4 | 2 | 7
Not completed — Lost to Follow-up | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone | Total
Number analyzed (Participants) | 16 | 15 | 14 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 15 | 14 | 45
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 6 | 19
  Male | 7 | 11 | 8 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome as Measured in Length of Time to Meet Return To Sport Criteria (Measured in Days)
Description: The Return To Sport Criteria is met when all items on the Return To Sport Checklist can be successfully achieved. There are no units of measure for any of the criteria listed as they are either achieved/passed or not achieved/failed based on the criteria listed. Once all criteria can be passed, this date is noted. The number of days from Visit 1 to the date when all criteria are achieved is calculated. This outcome is measured in days.
Time Frame: Measured at each Study Treatment Visit for a maximum of 12 Study Treatment Visits over a maximum of 8 weeks or until Return to Sport Criteria are met, whichever is sooner
Population: Analysis of return to sport time in patients who met return to sport criteria during study
Measure: Mean (Standard Deviation); unit: days to meet return to sport criteria
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
Number analyzed (Participants) | 7 | 9 | 4
days to meet return to sport criteria | 38.1 (9.48) | 30.2 (6.8) | 37.25 (3.86)
Statistical Analysis 1: Comparison: Iontophoresis With Dexamethasone vs Iontophoresis With Sodium Chloride; Test type: Equivalence — p<0.05 was considered statistically significant. A 95% confidence interval was computed using logistic regression model; p = 0.0366, Cox proportional hazards analysis; Hazard Ratio (HR) = 3.11, 95% CI 2-sided [1.073 to 9.005]
Statistical Analysis 2: Comparison: Iontophoresis With Sodium Chloride vs Physical Therapy Alone; Test type: Equivalence — p<0.05 was considered statistically significant; p = 0.0232, Cox proportional hazards analysis; Hazard Ratio (HR) = 4.16, 95% CI 2-sided [1.215 to 14.273]
Statistical Analysis 3: Comparison: Iontophoresis With Dexamethasone vs Physical Therapy Alone; Test type: Equivalence — p<0.05 was considered statistically significant; p = 0.64, Cox proportional hazards analysis; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.389 to 4.615]

2. Secondary Outcome: Patient Reported Outcome - Percent Difficulty With Activities as Measured by the Lower Extremity Function Scale (LEFS)
Description: The LEFS is a patient reported questionnaire that measures difficult of completing 20 activities. The maximum possible score of the LEFS is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function. The LEFS data is reported as a percentage, calculated as XX points/80 * 100.
Time Frame: Collected at final visit, which is at Visit 12, maximum of 8 weeks, or when Return to Sport Criteria are met, whichever is sooner
Population: Analysis of final LEFS scores available across each group that completed full study participation. There were a total of 18 participants that did not complete their final LEFS scores across all three groups, so these patients have no final LEFS scores available for final analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
Number analyzed (Participants) | 8 | 11 | 8
percent | 84.66 (17.50) | 86.42 (12.89) | 81.98 (23.38)
Statistical Analysis 1: Comparison: Iontophoresis With Dexamethasone vs Iontophoresis With Sodium Chloride vs Physical Therapy Alone; Test type: Equivalence — All statistical tests were two-sided, and p<0.05 was considered statistically significant; p = 0.86, ANOVA

3. Secondary Outcome: Patient Reported Outcome - Activity Level as Measured by the Godin Leisure-Time Activity Questionnaire
Description: The Godin Leisure-Time Activity Questionnaire measures physical activity. Scores of 24 and above indicate the individual is "Active", scores of 14-23 indicate the individual is "Moderately Active", and scores of 14 and below indicate the individual is insufficiently active/sedentary. A higher score indicates higher levels of physical activity at baseline, thus would be considered a better outcome. The minimum possible score is 0, and there is no defined maximum score, as scores are based on patient's self-reported quantitative activity level, but scores of 24 and above indicate the highest levels of physical activity.
Time Frame: Measured at Study Treatment Visit 1 to establish baseline activity level (prior to onset of injury/pain)
Population: Analysis of initial Godin scores between groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
Number analyzed (Participants) | 16 | 15 | 14
score on a scale | 71.81 (23.61) | 58.07 (24.86) | 65.43 (18.54)
Statistical Analysis 1: Comparison: Iontophoresis With Dexamethasone vs Iontophoresis With Sodium Chloride vs Physical Therapy Alone; Test type: Equivalence — p<00.05 was considered statistically significant; p = 0.25, ANOVA

4. Secondary Outcome: Patient Reported Outcome - Pain as Measured by the Wong-Baker FACES Pain Rating Scale
Description: This scale was created for children to help them communicate their pain. The scale shows a series of faces ranging from a happy face at 0, "No hurt" to a crying face at 10 "Hurts worst".
Time Frame: as for outcome 2
Population: Analysis of final FACES Pain scale ratings across all groups as available. We had 13 patients who did not provide final FACES pain data, thus that data was unable to be included in final analysis.
Measure: Mean (Standard Deviation); unit: score on a scale of 0-10
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
Number analyzed (Participants) | 11 | 12 | 10
score on a scale of 0-10 | 1.33 (0.65) | 1.85 (1.07) | 2.13 (1.36)
Statistical Analysis 1: Comparison: Iontophoresis With Dexamethasone vs Iontophoresis With Sodium Chloride vs Physical Therapy Alone; Test type: Equivalence — p<0.05 considered statistically significant; p = 0.29, ANOVA

5. Secondary Outcome: Number of Participants With Adverse Events
Description: All adverse events that occur during participation in this research study, whether or not considered intervention-related, will be collected.
Time Frame: Measured at each Study Treatment Visit (up to 12 Study Treatment Visits over a maximum of 8 weeks or until Return to Sport Criteria are met, whichever is sooner), then again 2 - 3 days, 30 days, and 90 days after Return To Sport Criteria are met.
Population: Participants in each group who experienced an AE
Measure: Count of Participants; unit: Participants
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
Number analyzed (Participants) | 14 | 10 | 9
Participants
  Mild AE | 8 | 5 | 4
  Moderate | 4 | 5 | 5
  Severe | 2 | 0 | 0
Statistical Analysis 1: Comparison: Iontophoresis With Dexamethasone vs Iontophoresis With Sodium Chloride vs Physical Therapy Alone; Test type: Equivalence — All statistical tests were performed using the SAS Studio. All statistical tests were two-sided, and p<0.05 was considered statistically significant; p = 0.57, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were tracked throughout the study duration for each participant, i.e. approximately 5 months.
Arm/Group | Iontophoresis With Dexamethasone | Iontophoresis With Sodium Chloride | Physical Therapy Alone
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 14/16 | 10/15 | 9/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iontophoresis With Dexamethasone (N=16) | Iontophoresis With Sodium Chloride (N=15) | Physical Therapy Alone (N=14)
lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — 1 1/2 cm x 3 1/2 cm lesion
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — to right knee
bilateral foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
bruised elbow (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
common cold (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
concussion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
fractured clavicle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
left arm soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
patellar tendinopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
redness at patch site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
redness superior to patch location (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
anterior knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
foot/great toe pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
knee pain with flexion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
tibial tubercle hyperpigmentation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
tibial tubercle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
rolled ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
small red bumps around tibia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
bruising around patch area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
dryness over tibial tubercle (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
pressure sensation under patch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
stinging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Our study was limited by limited enrollment, primarily as a result of the COVID-19 pandemic. Slow enrollment following the pandemic led to early closure of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03606980/Prot_SAP_000.pdf